CLINICAL TRIAL: NCT02151097
Title: A Feasibility Study to Evaluate 18F-choline Cerenkov Luminescence Imaging for Measuring Margin Status in Radical Prostatectomy Specimens
Brief Title: PRIME - PRostate Imaging for Margin Evaluation
Acronym: PRIME
Status: Completed | Type: Observational
Sponsor: Lightpoint Medical Limited (Industry)
Collaborators: University College London Hospitals (Other); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: LPM-003
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-03

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatectomy; Prostate cancer; Cerenkov Luminescence Imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High risk prostate cancer: Men ≥18 years of age diagnosed with high risk prostate cancer, defined as clinical stage ≥T2c, or Prostate Specific Antigen (PSA)>20 ng/ml, or Gleason Score 8-10, scheduled to have radical prostatectomy.

SUMMARY:
This study will evaluate the feasibility of using intra-operative Cerenkov Luminescence Imaging (CLI) of prostatectomy specimens to determine tumour margin status. The samples will be imaged using the LightPathTM Imaging System which consists of a light-tight box containing an ultra-sensitive lens and radiation-shielded camera. This study will measure the correlation between margin status of the WLE specimen and the metastatic status of dissected lymph nodes as determined by the LightPathTM Imaging System and by histopathology. This is a pilot study to assess feasibility before proceeding to a pivotal study to evaluate the benefits of the LightPathTM system in clinical practice.

DETAILED DESCRIPTION:
This study is a prospective, single-centre feasibility study to evaluate the use of intra-operative Cerenkov Luminescence Imaging (CLI) of prostatectomy specimens to determine margin status.

Subjects will receive an intravenous injection of 370 Mega Becquerel (MBq) of 18F-choline prior to routine, elective radical prostatectomy. The surgery will be performed according to standard-of-care. The resected prostatectomy specimens will be imaged using the LightPathTM Imaging System, consisting of a light-tight box containing an ultra-sensitive lens and Electron Multiplying Charged-Coupled Device (EMCCD) camera.

This study will measure the agreement between margin status of the prostatectomy specimen as determined by CLI and by histopathology (reference method). This study will assess feasibility before proceeding to a pivotal study to evaluate the benefits of the LightPathTM Imaging System in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥18 years of age diagnosed with high risk prostate cancer, defined as clinical stage ≥T2c, or PSA>20 ng/ml, or Gleason Score 8-10.
* Patients undergoing radical prostatectomy

Exclusion Criteria:

* Known hypersensitivity to 18F-choline
* Patients currently taking colchicine
* Prior therapy for prostate cancer (e.g. focal therapy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men ≥18 years of age diagnosed with high risk prostate cancer, defined as clinical stage ≥T2c, or PSA>20 ng/ml, or Gleason Score 8-10, undergoing radical prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Margin status of prostatectomy specimen as determined by the LightPathTM Imaging System | Intra-operative
  Use of the LightPathTM Imaging System will be examined in order to assess the feasibility of using CLI for determining margin status intraoperatively.

SECONDARY OUTCOMES:
The agreement between margin status as determined by CLI and histopathology | Intra and immediate post-operative
  Tumour margin status of prostatectomy specimens as determined by CLI and routine histopathology analysis will be compared in order to assess the performance of the LightPathTM Imaging System for determining margin status intraoperatively.

OTHER OUTCOMES:
Radiation dosimetry to staff | Intra and immediate post-operative
  Radiation dosimetry results will be used to assess the feasibility of following routine procedures for care of patients and handling of surgical specimens in patients undergoing prostatectomy following administration of 18F-choline.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl O'Farrell, PhD, Study Director — Head of Clinical Development, Lightpoint Medical
Locations (1):
- University College Hospital London, London, United Kingdom